CLINICAL TRIAL: NCT07158164
Title: DPYD Pharmacogenomics and Fluoropyrimidine (FP) Dose-Adjustment
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Howard S. Hochster, MD, Distinguished Professor of Medicine, Director Clinical Oncology Research, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 072504
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Neoplasms; Breast Neoplasms; Head and Neck Neoplasms; Gastro-Intestinal Intraepithelial Neoplasia
Keywords: colorectal cancer; breast cancer; head and neck cancer; Gastro-Intestinal cancer; chemotherapy toxicity
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Head and Neck Neoplasms | interventions — Fluorouracil; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Normal DPYD Patients (Control Arm) (Active Comparator): Should receive 100% of the standard recommended doses as per the BEACON order plan.
  Dose Reduction for Toxicity: Reduce doses by 25% for unacceptable Grade 3 or any Grade 4 toxicity or clinically significant laboratory anbormaillity. If this occurs again, an additional 25% reduction (to 50% of the initial doses) should be used.
  Interventions: Drug: Fluorouracil injection; Drug: Xeloda
- Patients with One DPYD Variant (Heterozygotes) (Experimental): Will receive 50% of the regular starting doses for the first two cycles. For example, for FOLFOX or FOLFIRI, the 5FU bolus would be 200 mg/m², and the infusion would be 46 hours at 1200 mg/m².
  Interventions: Drug: Fluorouracil injection; Drug: Xeloda

INTERVENTIONS:
Drug: Fluorouracil injection — Experimental arm Fluorouracil injection with possible escalation to 75 or 100 percent if tolerated.
Drug: Xeloda — Experimental arm Fluorouracil injection with possible escalation to 75 or 100 percent if tolerated.

SUMMARY:
To prospectively evaluate the efficacy and safety of DPYD-guided dosing strategies in a real-world clinical setting, specifically by comparing the incidence of severe (Grade 3 and 4) fluoropyrimidine-related toxicities of heterozygous DPYD variant patients assigned to DPYD-guided reduced dosing versus patients with standard dosing in the control arm.

DETAILED DESCRIPTION:
Fluropyrimidines (FPs), such as 5-Fluorouracil (5-FU) and Capecitabine, are cornerstone chemotherapy agents widely used in the treatment of various cancers, including gastrointestinal, head and neck, and breast cancers. Dosing of FP, specifically 5-FU, has been a challenge since this drug was first synthesized in 1957 by Charles Heidelberger1. 5FU had been given on numerous schedules and doses, including weekly 24 hr infusion, 48-hour infusion every two weeks, and daily five-times-a-day infusion with leucovorin (Mayo Regimen) and weekly bolus with leucovorin infusion (Roswell, Park Regimen). In addition, oral fluropyrimidines, including Capecitabine, Tegafur, and S-1, are widely used throughout the world and have more prolonged dosing schedules, typically consisting of 2- to 3-week courses given twice daily. Despite their efficacy, the administration of these therapies has historically been challenging due to significant inter-patient variability in toxicity. A small but critical proportion of patients experience severe, potentially fatal toxicities, primarily attributed to a deficiency in Dihydropyrimidine Dehydrogenase (DPD) enzyme.

DPD is the key enzyme in the catabolism of 5-FU, metabolizing it into less toxic metabolites, such as FBAL. DPD activity may also be involved in decreasing the absorption of 5FU from the oral GI tract and accounts for its variability in absorption. When using irreversible DPD inhibitors, such as ethinyl-uracil, the daily oral dose of 5FU was less than 2 mg/m² compared to more than 1000 mg/m² when given orally.

Genetic variants in the DPYD gene, which encodes the DPD enzyme, are responsible for reduced or absent enzyme function. These variants are catalogued by the Clinical Pharmacogenetics Implementation Consortium (CPIC) and range from no function to reduced or normal function. While the prevalence of any DPYD reduced activity variant is estimated at 2-4% in the American population (heterozygous abnormality), homozygous abnormalities are much rarer (<0.0025%).

Historically, routine DPYD gene testing has not been widely recommended in the United States due to concerns about cost, treatment delays, and inconvenience2. However, the European community, with a higher incidence of DPYD deficiency and more affordable testing, has recommended routine testing for some time. However, the FDA only recently added a black box warning against using 5-FU in patients with DPD enzyme deficiency. On January 24, 2025, the FDA, as part of Project Renewal, recommended that clinicians consider testing all patients and discuss the issue with them. The FDA notes that for complete DPD deficiency, no dose is considered safe; however, for "partial deficiency," they state, "there is insufficient data to recommend a specific dose in patients with partial DPD deficiency."4

Given that the new warnings are now part of the package insert for 5-FU and Capecitabine, it is more incumbent on the practitioner to test for this abnormality for all patients beginning fluoropyrimidine therapy. CPIC has proposed reduction guidelines for patients with one gene abnormality (heterozygotes), which include a 50% dose reduction or possibly a 30% dose reduction for those with less severe DPD activity.³ However, these guidelines lack widespread clinical validation, raising questions about their necessity for toxicity control versus potential underdosing of such patients, affecting therapeutic outcomes. This prospective interventional treatment study aims to validate these DPYD-guided dosing strategies in a real-world clinical setting

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer in either the adjuvant or metastatic setting requiring initial therapy with 5-FU or Capecitabine.
* DPYD testing performed by a CLIA-certified laboratory (i.e., Guardant 360 or Caris blood testing for genomic profiling, DPYD testing by the Mayo Clinic or other certified laboratory) with results available before starting chemotherapy.
* DPYD testing results falling into one of the following cohorts for first-line therapy with a fluoropyridine:
* Study Cohort: Patients with one DPYD variant in one gene (heterozygotes).
* Control Arm: Patients with normal or wild-type DPYD genes, for comparison, will be treated at the usual 100% dose.

  --FOLFOX regimen (N=50)
* ECOG Performance Status 0-2.
* Measurable disease or non-measurable disease allowed, including adjuvant 5-FU-based regimens.

Exclusion Criteria:

* Patients for whom 5-FU or Capecitabine therapy is contraindicated or not deemed appropriate in the judgment of the treating physician.
* Patients with two DPYD variants (homozygous deletions or non-functional genetic variants, or double heterozygotes with two different abnormalities) should not receive 5-FU or Capecitabine and are therefore excluded from the study.
* Pregnant Women and Children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2027-07-07 (Estimated); Study Completion 2029-07-07 (Estimated)

PRIMARY OUTCOMES:
incidence of severe fluoropyrimidine-related toxicities (Grade 3-5) | up to 24 months
  Number and proportion of patients experiencing Grade 3, 4, or 5 toxicities related to 5-FU or Capecitabine, as defined by CTCAE v5.0.

SECONDARY OUTCOMES:
Patterns of Dose Modification (Reductions and Escalations) | up to 24 months
  Number and type of dose modifications (reductions, escalations, discontinuations) in each arm,

CONTACTS AND LOCATIONS:
Overall Officials: Howard S. Hochster, MD, Principal Investigator — Study Principal Investigator
Locations (12):
- United States (12):
  - RWJBarnabas Health Clara Maas Medical Center, Belleville, New Jersey
  - Trinitas Hospital and Comprehensive Cancer Center, Elizabeth, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, Hamilton, Hamilton, New Jersey
  - RWJBarnabas Health Jersey City Medical Center, Jersey City, New Jersey
  - Cooperman Barnabas Medical Center, Livingston, New Jersey
  - Jack and Sheryl Morris Cancer Center, New Brunswick, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospita, New Brunswick, New Jersey
  - Cancer Center Initiative, Newark, New Jersey
  - University Hospital, Newark, New Jersey
  - RWJBarnabas Health Newark Beth Israel Medical Center, Newark, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - RWJBarnabas Health - Community Medical Center, Toms River, New Jersey

IPD SHARING:
Plan to Share IPD: No